CLINICAL TRIAL: NCT04737538
Title: A Randomized Controlled Examiner-blind Phase ii Proof-of-principle Clinical Study Investigating the Efficacy of an Experimental Dentifrice Containing Sodium Bicarbonate, High Molecular Weight Sodium Hyaluronate and Sodium Fluoride on Gingivitis and Plaque Removal in a Population With Mild-moderate Plaque-induced Gingivitis
Brief Title: A Proof-of-principle Clinical Study Investigating the Efficacy of an Experimental Dentifrice Containing Sodium Bicarbonate and Sodium Hyaluronate on Gingivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 208175
Record Dates: First submitted 2021-01-18; First posted 2021-02-04 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Dentifrice (Experimental): Participants assigned to this arm will apply full ribbon of toothpaste (containing sodium bicarbonate, sodium hyaluronate and sodium fluoride) to cover the head of toothbrush provided and will brush their teeth for one timed minute twice a day (morning and evening).
  Interventions: Other: Experimental Dentrifrice
- Positive control (Active Comparator): Participants assigned to this arm will apply full ribbon of toothpaste (dentifrice containing 67% w/w sodium bicarbonate and 0.221% w/w sodium fluoride) to cover the head of toothbrush provided and will brush their teeth for one timed minute twice a day (morning and evening).
  Interventions: Other: Positive control dentifrice
- Negative control (Active Comparator): Participants assigned to this arm will apply full ribbon of toothpaste (dentifrice containing 1100ppm fluoride as sodium fluoride [Crest Cavity Protection]) to cover the head of toothbrush provided and will brush their teeth for one timed minute twice a day (morning and evening).
  Interventions: Other: Negative control dentifrice

INTERVENTIONS:
Other: Experimental Dentrifrice — Toothpaste containing sodium bicarbonate, sodium hyaluronate and sodium fluoride
  Arms: Experimental Dentifrice
Other: Positive control dentifrice — Dentifrice containing 67% w/w sodium bicarbonate and 0.221% w/w sodium fluoride
  Arms: Positive control
Other: Negative control dentifrice — Dentifrice containing 1100ppm fluoride as sodium fluoride (Crest Cavity Protection)
  Arms: Negative control

SUMMARY:
The aim of this study is to develop a daily use toothpaste containing sodium bicarbonate, sodium hyaluronate and sodium fluoride with the intention of providing improved/ fast gum healing. This Proof-of-Principle study will investigate the efficacy of an experimental dentifrice compared to a regular fluoride dentifrice, and also whether this provides any additional benefit in reducing gingival inflammation/ bleeding compared with a 67% w/w sodium bicarbonate/ 0.221% w/w sodium fluoride containing toothpaste.

DETAILED DESCRIPTION:
This study will be a single-center, examiner-blind, randomized, stratified, three-treatment, parallel group study in healthy adult volunteers with mild to moderate gingivitis. There will be six visits to the study site: Screening, Baseline, Day 3 and Weeks 1, 2 and 6. Gingivitis will be assessed using a Modified Gingival Index (MGI) and a Bleeding Index (BI). Plaque will be assessed by the Turesky modification of the Quigley Hein (TPI). All evaluable teeth (in relation to the inclusion/ exclusion general dentition criteria) will be assessed.

The dosage regimen of twice daily treatment (morning and evening) for the washout dentifrice and study products will be the same for all participants and is based on widely recommended oral hygiene practice/typical consumer habit. Study participants will be instructed to brush for at least 1 timed minute with their assigned study dentifrice on each brushing occasion. After 6 weeks (Day 42+/-3 days) twice daily treatment, each participant should complete between approximately 84-90 treatment applications. During the washout period for this study (minimum 14 days/ maximum 28 days), eligible participants will use a marketed, regular fluoride toothpaste and toothbrush (as provided).

ELIGIBILITY:
Inclusion Criteria-

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant/relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Female participant of childbearing potential must have negative pregnancy test results at screening and baseline.
* Female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for 5 days after the last dose of assigned treatment. A female participant who is of childbearing potential must agree to use a highly effective method of contraception consistently and correctly for the duration of the active study period and for at least 5 days after the last dose of investigational product..

At Screening (Visit 1):

1. Participant with at least 20 natural, permanent teeth.
2. Participant with at least 40 evaluable surfaces for MGI, BI and TPI. An evaluable surface is defined as having 2/3rds of the natural tooth surface gradable for the selected clinical indices. The following should not be included in the evaluable surface count- third molars; fully crowned/extensively restored, grossly carious, orthodontically banded/bonded or abutment teeth; surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with the baseline assessments of the selected clinical indices.
3. Participant with generalized mild- moderate plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by a gross visual examination at the Screening Visit.

At Baseline - Prior to Dental Prophylaxis (Visit 2):

1. Participant with ongoing hard tissue eligibility and, in the opinion of the clinical examiner, at least 40 evaluable surfaces.
2. Participant with mean whole mouth MGI between 1.75 and 2.30.
3. Participant with mean whole mouth TPI score ≥1.5.
4. Participant with a minimum of 20 bleeding sites.

   Exclusion Criteria-
   * Participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GlaxoSmithKline Consumer Healthcare (GSKCH) employee directly involved in the conduct of the study or a member of their immediate family.
   * Participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
   * Participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee would make the participant inappropriate for entry into this study.
   * Participant with any other clinical serious or unstable conditions (e.g. cardiovascular diseases, diabetes, liver disorders and kidney disorders) which may affect study outcomes and/ or participant safety.
   * Participant who is a pregnant female (including a woman who has a positive urine pregnancy test; pregnancy testing will be carried out for all female participants who are of childbearing potential) or is intending to become pregnant over the duration of the study.
   * Participant who is a breastfeeding female.
   * Participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
   * Participant unwilling or unable to comply with the Lifestyle Considerations described below:

     1. Dental Product/Treatment and Oral Hygiene Restrictions From Screening (Visit 1) to the Participant's Last Study Visit • Participants should not use any other oral care products (e.g. dentifrices, toothbrushes, mouthrinses) other than those provided during the study.

        • Participants should not carry out any interproximal dental cleaning. Use of dental floss, toothpicks, waterpicks or inter-dental brushes is prohibited (except for the removal of impacted food with non-antimicrobial products only).

        • Participants should delay any non-emergency dental treatment until after study completion (including dental prophylaxis).

        Before Clinical Efficacy Assessment Visits: Baseline (Visit 2) to Last Study Visit • Participants should refrain from oral hygiene procedures for 12 hours ((+6hr, -2hr) before their visit and attend the study site with overnight plaque growth.
     2. Dietary and Smoking Restrictions From Screening (Visit 1) to the Participant's Last Study Visit • Participants should not chew gum or consume any confectionery containing xylitol (e.g. mints).

        * Participants must abstain from smoking/ use of tobacco products (e.g. chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).

   Before Clinical Efficacy Assessment Visits: Baseline (Visit 2) to Last Study Visit

   • Participants must abstain from all food and drink (except water) for at least 4hrs prior to their scheduled assessment visits and until all assessments are complete during visit days. Water is permitted until 1 hour prior to their scheduled study visits.

   - Participant who is a current smoker or an ex- smoker who stopped within 6 months of Screening.

   - Participant who currently uses smokeless forms of tobacco (e.g. chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).

   - Participant with diagnosed xerostomia or taking any medication that in the view of the investigator causes xerostomia.

   - Participant with a medical condition which may directly influence gingival bleeding.
   * Participant with a bleeding disorder that may affect study outcomes and/ or participant safety.
   * Recent history (within the last year) of alcohol or other substance abuse.
   * Participant with a severe oral condition (e.g. acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that would, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/ examiner if they were to participate in the study.
   * Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
   * Medication Exclusions

   At Screening (Visit 1):

<!-- -->

1. Participant currently taking antibiotics or requiring antibiotic use prior to dental prophylaxis or other dental procedures.
2. Participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
3. Participant currently taking a systemic medication (e.g. anti-inflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (e.g. ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).

   - Medication exclusions

   At Baseline (Visit 2):

<!-- -->

1. Participant who has taken (in the previous 14 days), any antibiotics.
2. Participant who has taken (in the previous 14 days) a systemic medication (e.g. antiinflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (e.g. ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
3. Participant who has used an antibacterial dentifrice or mouthwash (e.g. chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, in the period between Screening and the Baseline

   - Periodontal Exclusions

a. Participant with signs of active periodontitis. b. Participant with gingivitis which, in the opinion of the investigator, is not expected to respond to treatment with an over-the-counter dentifrice.

c. Participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.

* Dental Exclusions

  1. Participant with active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they were to participate in the study.
  2. Participant with dentures (partial or full).
  3. Participant with an orthodontic appliance (bands, appliances or fixed/ removable retainers).
  4. Participant who has received orthodontic therapy within 12 months of Screening.
  5. Participant with numerous restorations in a poor state of repair.
  6. Participant with any dental condition (e.g. overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they were to participate in the study.
  7. Participant who has had dental prophylaxis within 12 weeks of Screening.
  8. Participant who has had teeth bleaching within 12 weeks of Screening.
  9. Participant with high levels of extrinsic stain or calculus deposits that might interfere with plaque assessments.
* Participant who has previously been enrolled in this study.
* Participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be grant-ed, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Axe A, Patel N, Qaqish J, Ling MR, Araga M, Parkinson C, Goyal CR. Efficacy of an experimental toothpaste containing sodium bicarbonate, sodium hyaluronate and sodium fluoride on gingivitis. BMC Oral Health. 2024 Feb 9;24(1):209. doi: 10.1186/s12903-024-03981-9. PMID 38336635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in Canada.
Pre-assignment Details: A total of 110 participants were enrolled into the study and allocated to a randomized treatment. Of these 36 participants were randomized to the experimental dentifrice group and positive control dentifrice group each and 38 participants were randomized to the negative control dentifrice group. All the randomized participants completed the study.
Groups:
- Experimental Dentifrice: Participants were instructed to apply full ribbon of toothpaste (containing 67 percent [%] weight/weight [w/w] sodium bicarbonate, 0.2% w/w sodium hyaluronate and 0.221% w/w sodium fluoride) to cover the head of toothbrush provided and to brush their teeth for one timed minute twice a day (morning and evening) for 6 weeks.
- Positive Control Dentifrice: Participants were instructed to apply full ribbon of toothpaste (dentifrice containing 67% w/w sodium bicarbonate and 0.221% w/w sodium fluoride) to cover the head of toothbrush provided and to brush their teeth for one timed minute twice a day (morning and evening) for 6 weeks.
- Negative Control Dentifrice: Participants were instructed to apply full ribbon of toothpaste (dentifrice containing 0.221% w/w fluoride as sodium fluoride [Crest Cavity Protection]) to cover the head of toothbrush provided and to brush their teeth for one timed minute twice a day (morning and evening) for 6 weeks.
Period: Overall Study
Arm/Group | Experimental Dentifrice | Positive Control Dentifrice | Negative Control Dentifrice
Started | 36 | 36 | 38
Completed | 36 | 36 | 38
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: Comprised of all randomized participants who received at least one dose of the study product.
Groups:
- Experimental Dentifrice: Participants were instructed to apply full ribbon of toothpaste (containing 67% w/w sodium bicarbonate, 0.2% w/w sodium hyaluronate and 0.221% w/w sodium fluoride) to cover the head of toothbrush provided and to brush their teeth for one timed minute twice a day (morning and evening) for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Experimental Dentifrice | Positive Control Dentifrice | Negative Control Dentifrice | Total
Number analyzed (Participants) | 36 | 36 | 38 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.9 (14.49) | 41.5 (16.52) | 40.3 (13.41) | 39.9 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 22 | 66
  Male | 14 | 14 | 16 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 7 | 5 | 8 | 20
  Asian - Central/South Asian Heritage | 2 | 4 | 6 | 12
  Asian - East Asian Heritage | 0 | 0 | 5 | 5
  Asian - South-East Asian Heritage | 0 | 1 | 0 | 1
  White - Arabic/North African Heritage | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 25 | 24 | 19 | 68
  Multiple | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeding Sites at 6 Weeks (Comparison of Experimental Versus Negative Control Dentifrice)
Description: Number of bleeding sites were assessed by examiner by gently inserting a probe into the gingival crevice to a depth of approximately 1 millimeter (mm) and then running around the tooth (at an angle of approximately 60 degree to the long axis of the tooth), gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Gingival bleeding sites were assessed 30 seconds after probing. Analysis was performed using Analysis of Covariance (ANCOVA) model with study product group and gender as factors and baseline number of bleeding sites as covariate. The estimates were based on separate ANCOVA model using only the data for corresponding comparison (experimental dentifrice vs negative control dentifrice).
Time Frame: At Week 6
Population: Modified Intent-to-Treat (mITT) Population: Comprised of all randomized participants who received at least one dose of the study product and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Error); unit: Number of Sites
Arm/Group | Experimental Dentifrice | Negative Control Dentifrice
Number analyzed (Participants) | 36 | 38
Number of Sites | 9.5 (0.80) | 20.5 (0.78)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Negative Control Dentifrice; Test type: Other; p < 0.0001, Non-parametric method (Van Elteren test); Mean Difference (Final Values) = -11.0, 95% CI 2-sided [-13.3 to -8.8], Standard Error of Mean 1.12

2. Secondary Outcome: Number of Bleeding Sites at Week 6 (Comparison of Experimental Versus Positive Control Dentifrice)
Description: Number of bleeding sites were assessed by examiner by gently inserting a probe into the gingival crevice to a depth of approximately 1 mm and then running around the tooth (at an angle of approximately 60 degree to the long axis of the tooth), gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Gingival bleeding sites were assessed 30 seconds after probing. Analysis was performed using ANCOVA model with study product group and gender as factors and baseline number of bleeding sites as covariate. The estimates were based on separate ANCOVA model using only the data for corresponding comparison (experimental dentifrice vs positive control dentifrice).
Time Frame: At Week 6
Population: mITT Population
Measure: Mean (Standard Error); unit: Number of Sites
Arm/Group | Experimental Dentifrice | Positive Control Dentifrice
Number analyzed (Participants) | 36 | 36
Number of Sites | 9.8 (0.71) | 9.4 (0.71)
Statistical Analysis 1: Comparison: Experimental Dentifrice vs Positive Control Dentifrice; Test type: Other; p = 0.4488, Non-parametric method (Van Elteren test); Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.6 to 2.4], Standard Error of Mean 1.01

3. Secondary Outcome: Number of Bleeding Sites at Week 6 (Comparison of Positive Versus Negative Control Dentifrice)
Description: Number of bleeding sites were assessed by examiner by gently inserting a probe into the gingival crevice to a depth of approximately 1 mm and then running around the tooth (at an angle of approximately 60 degree to the long axis of the tooth), gently stretching the epithelium while sweeping from interproximal to interproximal along the sulcular epithelium. Gingival bleeding sites were assessed 30 seconds after probing. Analysis was performed using ANCOVA model with study product group and gender as factors and baseline number of bleeding sites as covariate. The estimates were based on separate ANCOVA model using only the data for corresponding comparison (positive control dentifrice vs negative control dentifrice).
Time Frame: At Week 6
Population: mITT Population
Measure: Mean (Standard Error); unit: Number of Sites
Arm/Group | Positive Control Dentifrice | Negative Control Dentifrice
Number analyzed (Participants) | 36 | 38
Number of Sites | 9.1 (0.85) | 20.6 (0.82)
Statistical Analysis 1: Comparison: Positive Control Dentifrice vs Negative Control Dentifrice; Test type: Other; p < 0.0001, Non-parametric method (Van Elteren test); Mean Difference (Final Values) = -11.5, 95% CI 2-sided [-13.8 to -9.1], Standard Error of Mean 1.18

ADVERSE EVENTS:
Time Frame: From screening up to Week 6, up to approximately 70 days
Description: Adverse events were to be collected for safety population which included all randomized participants who received at least one dose of study product. However no deaths, adverse events or serious adverse events were reported.
Arm/Group | Experimental Dentifrice | Positive Control Dentifrice | Negative Control Dentifrice
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT04737538/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/38/NCT04737538/SAP_001.pdf